CLINICAL TRIAL: NCT04666935
Title: The Effect of the Oslo Sports Trauma Research Center (OSTRC) Injury Prevention Exercises Reducing Injuries Rate Among Athletes. a Randomized Controlled Trial.
Brief Title: The Effect of the Oslo Sports Trauma Research Center (OSTRC) Injury Prevention Exercises Reducing Injuries Rate Among Athletes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Wesam Saleh A. Al Attar, PT, MSc, PhD, Professor, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HAPO-02-K-012-2020-10-465
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Sport Injury
Keywords: Oslo Sports Trauma Research Center; Injury Prevention Program

STUDY DESIGN:
Intervention Model Description: The intervention group will be instructed to include the Oslo Sports Trauma Research Center (OSTRC) Injury Prevention Program as a warm up before training session (3 times per week) during one season (6 months).The control group will practice their usual warm up.
  Usual warm up is defined as any basic exercises performed before a performance or practice to prepare the muscles for vigorous actions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will be instructed to include the Oslo Sports Trauma Research Center (OSTRC) Injury Prevention Program as a warm up before training session (3 times per week) during one season (6 months).
  Interventions: Other: The Oslo Sports Trauma Research Center (OSTRC) Injury Prevention Program
- Control group (Active Comparator): The control group will practice their usual warm up. Usual warm up is defined as any basic exercises performed before a performance or practice to prepare the muscles for vigorous actions.
  Interventions: Other: Usual warm up

INTERVENTIONS:
Other: The Oslo Sports Trauma Research Center (OSTRC) Injury Prevention Program — Sport Injury Prevention Program.
  Arms: Intervention group
Other: Usual warm up — Usual warm up is defined as any basic exercises performed before a performance or practice to prepare the muscles for vigorous actions.
  Arms: Control group

SUMMARY:
The Oslo Sports Trauma Research Center (OSTRC) was established in May 2000 at the Norwegian School of Sport Sciences.The OSTRC aims to prevent injuries and other health problems related to sports. The majority of the research conducted at OSTRC involves elite sports.

The purpose of this study is to investigate the effect of the Oslo Sports Trauma Research Center (OSTRC) Injury Prevention Program in reducing injuries among athletes.

Hypothesis: that Oslo Sports Trauma Research Center (OSTRC) Injury Prevention Program has a beneficial effect in terms of injury prevention.

The purpose of this study is to investigate the effect of the Oslo Sports Trauma Research Center (OSTRC) Injury Prevention Program in reducing injuries among athletes.

DETAILED DESCRIPTION:
Study type Interventional Description of intervention(s) / exposure: The intervention group will be instructed to include the Oslo Sports Trauma Research Center (OSTRC) Injury Prevention Program as a warm up before training session (3 times per week) during one season (6 months).

Group sessions will be administered by an exercise physiologist and/ or athletic trainer and/ or soccer coaches and/ or strength and conditioning specialists and/ or physiotherapist.

Session attendance checklists will be used to assess or monitor adherence to the intervention.

Comparator / control treatment The control group will practice their usual warm up.

Usual warm up is defined as any basic exercises performed before a performance or practice to prepare the muscles for vigorous actions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Amateur Athletes
* Training at least three times per week

Exclusion Criteria:

* History of lower extremity injury requiring medical attention in the past 6 months
* Systemic diseases
* Cardiovascular disease
* Neurological disorders
* Bone fractures
* Surgery in the previous year.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-01-16 (Estimated); Primary Completion 2021-01-16 (Estimated); Study Completion 2021-06-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of initial injuries. | At the end of the intervention season (6 months).
  Injury is defined according to a consensus statement on injury definitions and data collection procedures in soccer studies; an injury will be recorded if it caused the player to be unable to completely participate in the following match or training session.Injury rates will be summarised as number of injuries per 1000 player-hours for both matches and training. Exposure time in hours will be calculated for each team over a 6-month period.
The incidence of recurrent injuries | At the end of the intervention season (6 months)
  Recurrent injury is defined as a repeat episode of a fully recovered injury. Injury is defined according to a consensus statement on injury definitions and data collection procedures in soccer studies; an injury will be recorded if it caused the player to be unable to completely participate in the following match or training session.

SECONDARY OUTCOMES:
injury severity | At time of any injury occurring throughout intervention soccer season (6 months)
  Defined as time loss in days (days unable to train): minor (1 to 7 days lost), moderate (8 to 21 days lost), or severe (>21 days lost). Injury severity data will be collected from Sports Injury Tracker injury reporting form.
Compliance with the intervention | At the end of the intervention season (6 months)
  the rate of compliance

CONTACTS AND LOCATIONS:
Locations (1):
- Umm Al Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Start: Immediately following publication. End: 5 years
Access Criteria: Access subject to approvals by Principal Investigator. The Principal Investigator can be contacted by email wsattar@uqu.edu.sa

REFERENCES:
- [Background] Al Attar WSA, Alshehri MA. A meta-analysis of meta-analyses of the effectiveness of FIFA injury prevention programs in soccer. Scand J Med Sci Sports. 2019 Dec;29(12):1846-1855. doi: 10.1111/sms.13535. Epub 2019 Sep 5. PMID 31394009
- [Background] Al Attar WSA, Soomro N, Pappas E, Sinclair PJ, Sanders RH. Adding a post-training FIFA 11+ exercise program to the pre-training FIFA 11+ injury prevention program reduces injury rates among male amateur soccer players: a cluster-randomised trial. J Physiother. 2017 Oct;63(4):235-242. doi: 10.1016/j.jphys.2017.08.004. Epub 2017 Sep 20. PMID 28939307
- [Background] Al Attar WS, Soomro N, Pappas E, Sinclair PJ, Sanders RH. How Effective are F-MARC Injury Prevention Programs for Soccer Players? A Systematic Review and Meta-Analysis. Sports Med. 2016 Feb;46(2):205-17. doi: 10.1007/s40279-015-0404-x. PMID 26403470